CLINICAL TRIAL: NCT00208650
Title: Non-Invasive Quantitation of Myocardial Dysfunction by Tissue Doppler/Synchronization Imaging After Orthotopic Heart Transplantation in Children
Brief Title: Tissue Doppler Echo Imaging of Heart Function After Transplant
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, William T. Mahle, MD, Principal Investigator, Emory University
Other Study IDs: 0620-2004
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Children With Heart Transplants
Keywords: pediatrics; transplant; cardiac

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
There are many children born with Congenital Heart Disease. Many of these children have to undergo surgical procedures to correct the problem. Some patients must eventually get a new heart. Once they get a new heart, we have to have ways to determine how well the new heart is doing inside of the body. Tissue Doppler Imaging is one way of doing so. Tissue Doppler Imaging is like an ultrasounds. It takes pictures of the heart. In addition to Tissue Doppler Imaging, there is a newer non-invasive procedure called Tissue Synchronization Imaging which will allow us to see how well the new heart is working as well. In this study we would use both techniques to determine how well the new heart is working.

DETAILED DESCRIPTION:
Heart transplantation is the only hope for children with end stage heart disease. Eventually cardiac deterioration occurs and leads to death or re-transplantation. Our understanding of the pathophysiology of cardiac dysfunction in these children is incomplete. The time course of the dysfunction process either in the RV and/or the LV, systole or diastole has never been studied in children. No meaningful TSI quantitation has ever been performed in a large pediatric OHT patient population. The long-term goal of this study will be the detection of functional myocardial changes associated with known stages post heart transplantation using TDI and TSI. These achievements impact the survival and quality of life of children after cardiac transplantation.

Research Design and Methods

All subjects who are treated in the transplant clinic will be approached for possible participation into the study. These patients will include newly transplanted (OHT) patients as well as patients who underwent OHT prior to the enrollment year. The following procedures will occur at each study visit:

Echocardiographic assessment Standard 2-dimensional, M-mode, and Doppler or 3-dimensional echocardiography evaluation will be performed. We will assess cardiac function using left ventricular shortening (SF) and ejection fractions (EF). The EF will be calculated using both M-Mode and by Simpson's rule. We will also perform tissue synchronization imaging (TSI) and tissue Doppler imaging (TDI) using the GE Vivid 7 echocardiographic system. Both TSI and TDI will assist investigators in assessing mechanical synchrony. In newly transplanted patients, these echocardiographic assessments will occur during the first 5 days to serially measure ventricular synchrony during the acute post-operative period. For older transplant patients and for new transplant patients greater than five days out from transplantation, echocardiographic studies will occur at all follow-up clinic visits as determined by physician preference.

Clinical assessment Clinical evaluation will be performed during all follow-up visits in order to track unrecognized complications or adverse events. As is standard, all patients undergoing transplantation follow-up will have an electrocardiogram (EKG) performed to assess rhythm.

ELIGIBILITY:
Inclusion Criteria:

- Children who have had cardiac transplant within one year.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75
Dates: Start 2005-09; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Fyfe, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States

REFERENCES:
- [Background] Boucek MM, Faro A, Novick RJ, Bennett LE, Keck BM, Hosenpud JD. The Registry of the International Society for Heart and Lung Transplantation: Fourth Official Pediatric Report--2000. J Heart Lung Transplant. 2001 Jan;20(1):39-52. doi: 10.1016/s1053-2498(00)00243-6. No abstract available. PMID 11166611
- [Background] Kanter KR, Tam VK, Vincent RN, Cuadrado AR, Raviele AA, Berg AM. Current results with pediatric heart transplantation. Ann Thorac Surg. 1999 Aug;68(2):527-30; discussion 530-1. doi: 10.1016/s0003-4975(99)00616-5. PMID 10475423